CLINICAL TRIAL: NCT02223793
Title: Effects of Cardiovascular Risk Screening in Pharmacies: A Randomized Study
Brief Title: Vascular Lifestyle-Intervention and Screening in Pharmacy
Acronym: VISA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oslo (Other)
Collaborators: University of Tromso (Other); University of Minnesota (Other); Boots Norway AS (Unknown); Mills DA (Industry)
Responsible Party: Principal Investigator, Karianne Svendsen, PHD student, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2013/1660; 39255 (NSD) (Registry Identifier: Norwegian Social Science Data Services); 1660/2013 (Registry Identifier: Regional committees for medical and health research ethics: South-East)
Record Dates: First submitted 2014-08-18; First posted 2014-08-22 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Diseases; Hypercholesterolemia; Dyslipidemia; Hypertensive Disease; Diabetes Mellitus, Type 2
Keywords: Vascular screening; Cardiovascular risk factors; Blood pressure; Lipids; Lifestyle; Identifying unknown risk; Low socioeconomic status; low threshold
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia; Dyslipidemias; Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- No information on high risk factor levels but lifestyle advice (Experimental): This arm of high risk participants will not be informed about their measured levels of the different cardiovascular risk factors at baseline. However, they will receive general information on how to lower risk factor levels in 8 weeks
  Interventions: Behavioral: No information on high risk factor levels but lifestyle advice
- No information on high risk factor levels nor lifestyle advice (Experimental): In this arm, participants will not be informed about their measured levels of the different cardiovascular risk factors, nor receiving lifestyle advices at baseline
  Interventions: Behavioral: No information on high risk factor levels, nor lifestyle advice
- Information on high risk factor levels and lifestyle advice (Experimental): This arm of high risk participants will not be informed about their measured levels of the different cardiovascular risk factors at baseline, and receive general information on how to lower risk factor levels in 8 weeks
  Interventions: Behavioral: Information on high risk factor levels and lifestyle advice

INTERVENTIONS:
Behavioral: Information on high risk factor levels and lifestyle advice — This arm of high risk participants will be informed about their measured levels of the different cardiovascular risk factors. They will also receive information on how to lower their levels in 8 weeks
  Arms: Information on high risk factor levels and lifestyle advice
Behavioral: No information on high risk factor levels but lifestyle advice — In this arm, participants will have delayed information on their risk factor levels, but they will receive general advices on how to lower levels in 8 weeks
  Arms: No information on high risk factor levels but lifestyle advice
Behavioral: No information on high risk factor levels, nor lifestyle advice — In this arm, participants will have delayed information on both their risk factor levels and general information on how to lower risk factor levels.
  Arms: No information on high risk factor levels nor lifestyle advice

SUMMARY:
The overall goal of the present project is to contribute to new knowledge about the effect of a low threshold population screening system for cardiovascular risk factors in Norway. Further, this project aim to study if identifying high cardiovascular risk itself may lead to beneficial changes in health behaviors such as physical activity, diet, tobacco and alcohol behavior together with reduced risk score of cardiovascular disease, across socioeconomic status. This fall, a nationwide, free screening of cardiovascular risk factors will be conducted in 150 pharmacies in Norway. All participants that consent to participate will measure full lipid-profile, blood pressure, HbA1c, body weight and height by health care providers in pharmacies. Based on their measurement levels, participants will be stratified into either a low or a high risk group. In the high risk group, participants will further be randomized to either the intervention group or one of the two control groups. Participants in the intervention group will be informed about all their measurement levels with comparison to the recommended levels. Contrary, participants randomized to the two control groups will have delayed information of their measured levels. Participants in the intervention group and the first control groups will receive general oral and written information about how to lower their measurement levels in 8 weeks. In the second control group, participants will not receive any information at the first visit. In this way the investigators may be able to isolate the effect of identifying high risk and high levels of the risk factors itself. All groups will be given a diet- and physical activity questionnaire at visit 1, and will be invited back after 8 weeks to once more perform the measurement screening and receive the same questionnaire. At visit 2, all participants will, after the measurement screening, be informed about their measured risk factors and receive information on how to lower their levels. 1 year after inclusion, all participants in the three groups will be invited back for a one-year follow up visit in pharmacy.

DETAILED DESCRIPTION:
One year after inclusion, all participants that were not loss to follow up, or had their consent withdrawn, were invited back to pharmacies to perform the same measurements for the third time. However, at this third visit, pharmacies were randomized 1:2 to test an additional intervention. Further, an extra blood sample, dried blood spot, was taken to measure cholesterol, HbA1c and fatty acids.

About half of the pharmacies (n=23) communicated cardiovasular disease (CVD) risk factor levels as Heart age compared to own age (British communication tool) together with tailored lifestyle advices on how to reduce elevated levels. While the other 25 pharmacies communicated CVD risk the usual way and gave general lifestyle advices on how to reduce CVD risk. 4 weeks later, all participants took dried blood spot samples at home. We will compare results from dried blood spot samples to study whether heart age and tailored lifestyle advice is more effective than general information in reducing CVD risk.

The investigators will also record social security number to make connection to central health registry as prescription registry, patient registry and cause of death registry after 2 years and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Above18 years
* Not pregnant or lactating
* Not previous cardiovascular events nor treatment related to cardiovascular disease ((myocardial infarction, stroke, angina pectoris, coronary artery bypass, - Percutaneous coronary intervention, diabetes type 1 and 2)
* No use of cholesterol lowering medication, bloodpressure lowering medication, bloodsugar lowering medication or medication related to diabetes

Exclusion Criteria:

* Below18 years
* Pregnant or lactating
* Previous cardiovascular events nor treatment related to cardiovascular disease (myocardial infarction, stroke, angina pectoris, coronary artery bypass,
* Percutaneous coronary intervention, diabetes type 1 and 2)
* Use of cholesterol lowering medication, bloodpressure lowering medication, bloodsugar lowering medication or medication related to diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2022-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Karianne Svendsen, M.Sc., Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, P.B. 1046 Blinderen, Norway

REFERENCES:
- [Derived] Svendsen K, Telle-Hansen VH, Morch-Reiersen LT, Garstad KW, Thyholt K, Granlund L, Henriksen HB, Gran JM, Jacobs DR Jr, Retterstol K. A randomized controlled trial in Norwegian pharmacies on effects of risk alert and advice in people with elevated cardiovascular risk. Prev Med Rep. 2018 Aug 9;12:79-86. doi: 10.1016/j.pmedr.2018.08.004. eCollection 2018 Dec. PMID 30191097

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Information on High Risk Factor Levels But Lifestyle Advice | No Information on High Risk Factor Levels Nor Lifestyle Advice | Information on High Risk Factor Levels and Lifestyle Advice
Started | 185 | 199 | 198
Completed | 168 | 190 | 185
Not Completed | 17 | 9 | 13
Not completed — Lost to Follow-up | 10 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 2 | 3
Not completed — Moved/studycenter unable to participate | 4 | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Information on High Risk Factor Levels But Lifestyle Advice | No Information on High Risk Factor Levels Nor Lifestyle Advice | Information on High Risk Factor Levels and Lifestyle Advice | Total
Number analyzed (Participants) | 185 | 199 | 198 | 582
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 113 | 124 | 131 | 368
  >=65 years | 72 | 75 | 67 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (14.6) | 56.5 (15.5) | 55.7 (14.4) | 56.5 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 136 | 141 | 417
  Male | 45 | 63 | 57 | 165
Region of Enrollment [Number; unit: participants]
  Norway | 185 | 199 | 198 | 582
Ad hoc risk score [Mean (Standard Deviation); unit: units on a scale] — Ad hoc riskscore IS a summarization of scores ranging from zero (favorablemeasures) to four (very unfavorable measures), assigned for each of TC, HDL-C, HbA1c, blood pressure, BMI and age. A risk score of≥4 served as inclusion criteria because it indicated moderately elevated risk of CVD (minimum score). Maximum score was 14.
  units on a scale | 5.2 (1.3) | 5.4 (1.5) | 5.4 (1.5) | 5.3 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in ad Hoc Risk Score (Measure on a Scale From Min 4 to Max 14)
Description: The (ad hoc) risk score was a summarization of points ranging from 0 (favorable measures) , 2 (slighly unfavourable) or 4 (very unfavorable measures) assigned for each of Total cholesterol, HDL-cholesterol, HbA1c, blood pressure, body mass index and age (age was included because presence of elevated cardiovascular disease risk factors is more alarming in younger age).
  Risk points for each risk factor was summarized into an total risk score ranging from 4 (min) to 14 (max). A total risk score of ≥4 served as inclusion criteria because it indicated moderately elevated risk of cardiovascular disease.
Time Frame: Baseline and at 8 weeks
Population: Between groups analysis
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | No Information on High Risk Factor Levels But Lifestyle Advice | No Information on High Risk Factor Levels Nor Lifestyle Advice | Information on High Risk Factor Levels and Lifestyle Advice
Number analyzed (Participants) | 185 | 199 | 198
units on a scale | -0.71 [-0.99 to -0.44] | -0.76 [-1.02 to -0.5] | -0.36 [-0.62 to -0.09]

2. Secondary Outcome: 8-week Change in Total Cholesterol
Description: Change in total cholesterol, from date of randomization and until the end of the follow up after 8 weeks.
Time Frame: At baseline and at 8 weeks
Population: Difference between three groups.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | No Information on High Risk Factor Levels But Lifestyle Advice | No Information on High Risk Factor Levels Nor Lifestyle Advice | Information on High Risk Factor Levels and Lifestyle Advice
Number analyzed (Participants) | 168 | 190 | 185
mmol/L | -0.12 [-0.23 to -0.06] | -0.16 [-0.31 to -0.02] | -0.08 [-0.23 to 0.06]

3. Other Pre Specified Outcome: Effect of Heart Age and Tailord CVD Advice After 1 Year
Description: Comparing results from blood samples after 4 weeks in 23 pharmacies (enhanced CVD communication) versus 25 pharmacies (general communication of CVD risk).N
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2020-04

ADVERSE EVENTS:
Time Frame: Adverse effects were collected during the study periode (1 year and 2 months)- between start of study (september 2014) and end of study (november 2015).
Description: Definition do not differ. adverse event collection was non-systematically where the subjects were adviced to contact PI or study coordinator.
Arm/Group | No Information on High Risk Factor Levels But Lifestyle Advice | No Information on High Risk Factor Levels Nor Lifestyle Advice | Information on High Risk Factor Levels and Lifestyle Advice
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/199 | 0/198
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/199 | 0/198
Other Adverse Events (participants affected / at risk) | 0/185 | 0/199 | 0/198

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No